CLINICAL TRIAL: NCT03924921
Title: The Effectiveness of a Relaxation Technique on the Quality of Life and Symptoms in People Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016-5940:PRG
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-04

CONDITIONS: HIV
Keywords: relaxation; quality of life; symptoms; pain; depression; anxiety; sleep problems; fatigue
MeSH Terms: conditions — Pain; Depression; Anxiety Disorders; Parasomnias; Fatigue | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenic training (Experimental): Autogenic training
  Interventions: Other: autogenic training
- wait list (Experimental): usual care for 6 months Autogenic training after 6 months
  Interventions: Other: autogenic training

INTERVENTIONS:
Other: autogenic training — autogenic training

SUMMARY:
Quality of life of people living with HIV is strongly affected by the presence of one or more symptoms, such as sleep problems, fatigue, muscle pain, anxiety and depressive symptoms. Autogenic training has shown positive effects on these symptoms in different populations, but there is very little evidence on the effects of this relaxation technique in people living with HIV.

DETAILED DESCRIPTION:
The aim of this project is to evaluate the effectiveness of a relaxation technique, autogenic training, on the quality of life and the physical and psychological symptoms in people living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18 ;
* have a diagnosis of HIV;
* present at least one of the following symptoms during the preceding two weeks: sleep problems, fatigue, pain, anxiety or symptoms of depression;
* understand and speak French and;
* be able to follow the instructions to learn the relaxation technique.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Quality of Life-human immunodeficiency virus (PROQOL-HIV) | 3 and 6 months
  The PROQOL-HIV questionnaire is composed of 43 Likert-type items (5-point scale ranging from 0=never to 4=always), including 39 items targeting 8 domains of HRQL and general health: physical health and symptoms (9 items), treatment impact (10 items), emotional distress (4 items), health concerns (4 items), body change (4 items), intimate relationships (3 items), social relationships (2 items), and stigma (2 items). Four extra items dealing with religious beliefs, finance, having children, and satisfaction with care are not part of the scoring scheme, but are used to gather additional information from the respondent. Responses to items will be totaled for each dimension and standardized on a scale from 0 to 100 points, in which higher values indicate a better health state.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | 3 and 6 months
  Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality and quantity. The19-item self-report questionnaire yields 7 component scores: subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction each weighted equally on a 0-3 scale. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality.
Fatigue Severity Scale (FSS) | 3 and 6 months
  Fatigue severity scale (FSS) is a 9-items instrument with seven items related to fatigue interference, one item related to the experience of fatigue itself and one item about what causes fatigue. Each item is scored on a 7-point Likert scale ranging from 1 (''strongly disagree'') to 7 (''strongly agree''). The mean score of the 9 items is used to estimate fatigue severity.
Brief Pain Inventory | 3 and 6 months
  Brief Pain Inventory (BPI) is a two-factor instrument that measures pain severity and pain interference. The pain severity factor has four items, all rated on a 0 ''No pain'' to 10 ''Pain as bad as you can imagine'' Likert scale. The pain interference factor has seven items, all rated on a 0 ''Does not interfere'' to 10 ''Interferes completely'' Likert scale. Arithmetic mean of the four severity items can be used as measures of pain severity; the arithmetic mean of the seven interference items can be used as a measure of pain interference
State -Trait Anxiety Inventory (STAI) | 3 and 6 months
  State-Trait Anxiety Inventory (STAI) is a 40-items instrument that measures state anxiety and trait anxiety. Each type of anxiety has its own scale of 20 different questions that are scored on a 4-point Likert scale ranging from 1 "Almost never" to 4 "Almost always". Scores range from 20 to 80, with higher scores correlating with greater anxiety.
PHQ-9 | 3 and 6 months
  Patient Health Questionnaire (PHQ-9) is a 9-item instrument that measure depressive symptoms severity. PhQ-9 score ranges from 0 to 27, because each of the 9 items can be scores from 0 "not at all" to 3 "nearly every day". Higher scores indicate higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Ramirez-Garcia, PhD, Principal Investigator — Université de Montréal
Locations (2):
- Canada (2):
  - CHUM, Montreal, Quebec
  - CUSM, Montreal, Quebec